CLINICAL TRIAL: NCT05723549
Title: A Randomized, Open-label, Single-Dose, Parallel Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1803 in Healthy Male Volunteers.
Brief Title: A Study to Evaluate the PK, Safety and Tolerability of HCP1803.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-APOLLO-101
Record Dates: First submitted 2023-02-02; First posted 2023-02-10 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group1 (Experimental): Period1 : HCP1803-3
  Interventions: Drug: HCP1803-3
- group2 (Active Comparator): Period1 : RLD2002, HCP1904-1
  Interventions: Drug: RLD2002; Drug: HCP1904-1

INTERVENTIONS:
Drug: HCP1803-3 — Take it once per period
  Arms: group1
Drug: RLD2002 — Take it once per period
  Arms: group2
Drug: HCP1904-1 — Take it once per period
  Arms: group2

SUMMARY:
A randomized, open-label, single-dose parallel study to evaluate the pharmacokinetics, safety and tolerability of HCP1803 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy male volunteers
2. Weight ≥ 55kg and BMI 18 ~ 30 kg/m^2
3. Subjects who agree to use clinically accepted dual contraceptives up to 14 days after the last administration date of the investigational product and not to provide sperm.
4. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing.

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~144hours
  pharmacokinetic evaluation
AUC last | 0~144hours
  pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUC inf | 0~144hours
  pharmacokinetic evaluation
Tmax | 0~144hours
  pharmacokinetic evaluation
t1/2 | 0~144hours
  pharmacokinetic evaluation
CL/F | 0~144hours
  pharmacokinetic evaluation
Vd/F | 0~144hours
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No